CLINICAL TRIAL: NCT05292144
Title: Xperience Pro Post-Market Clinical Follow-up Study
Brief Title: Xperience Pro PMCF Study
Acronym: rEPIC04A
Status: Completed | Type: Observational
Sponsor: Fundación EPIC (Other)
Responsible Party: Sponsor
Other Study IDs: Xperience Pro PMCF Study
Record Dates: First submitted 2022-03-14; First posted 2022-03-23 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Coronary Artery Disease (CAD); Ischemic Heart Disease
Keywords: MDR (Medical Device Regulations); PMCF (Post-Market Clinical Follow-up); Coronary balloon dilatation catheter
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Coronary Artery Disease (CAD)
  Interventions: Device: Xperience Pro

INTERVENTIONS:
Device: Xperience Pro — Patients in whom treatment with (Xperience Pro) has been attempted

SUMMARY:
Multicenter, prospective, non-randomized, post-market clinical follow-up (PMCF) study to confirm and support the clinical safety and performance of Xperience Pro to meet EU Medical Device regulation (MDR) requirements in all the CONSECUTIVE patients treated with Xperience Pro .

DETAILED DESCRIPTION:
The objective of this multicenter, prospective, non-randomized, post-market clinical follow-up (PMCF) study is to confirm and support the clinical safety and performance of the Xperience Pro in a NON-SELECTED, Real World population under daily clinical practice when used as intended by the manufacturer to meet EU Medical Device regulation requirements for post-market clinical follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patient treated with Xperience pro according to routine hospital practice and following instructions for use
* Informed consent signed

Exclusion Criteria:

* Not meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with Xperience pro according to routine hospital practice and following instructions for use
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2022-10-26 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2023-05-05 (Actual)

PRIMARY OUTCOMES:
Safety Endpoint. Freedom from Target Lesion Failure | 7 days
  Freedom from TARGET LESION FAILURE (TLF), composite endpoint of cardiac death, myocardial infarction and and new Target Lesion Revascularization (TLR)

SECONDARY OUTCOMES:
Efficacy Endpoint. Freedom from Target Lesion Failure | 7 days
  Freedom from TARGET LESION FAILURE (TLF), composite endpoint of cardiac death, myocardial infarction (MI) and and new Target Lesion Revascularization (TLR).
Freedom from Balloon rupture | During percutaneous coronary intervention (PCI)
  Freedom from Balloon rupture
Freedom from Hypotube rupture | During PCI
  Freedom from Hypotube rupture
Freedom from Complicated withdrawal | During PCI
  Freedom from Complicated withdrawal
Freedom from Coronary perforation | During PCI
  Freedom from Coronary perforation
Freedom from Coronary dissection >C | During PCI
  Freedom from Coronary dissection >C
Freedom from No reflow | During PCI
  Freedom from No reflow
Freedom from Coronary thrombosis | During PCI
  Freedom from Coronary thrombosis

CONTACTS AND LOCATIONS:
Locations (5):
- Spain (5):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario de Getafe, Getafe
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Universitario Virgen de Valme, Seville

REFERENCES:
- [Background] Gruntzig A. Transluminal dilatation of coronary-artery stenosis. Lancet. 1978 Feb 4;1(8058):263. doi: 10.1016/s0140-6736(78)90500-7. No abstract available. PMID 74678
- [Background] Kandzari DE, Zankar AA, Teirstein PS, Brilakis ES, Banerjee S, Price MJ, Stinis CT, Hudson PA, Dahle TG, Eng M, Brown R, Ferguson A, Addo TA, Popma JJ. Clinical outcomes following predilation with a novel 1.25-mm diameter angioplasty catheter. Catheter Cardiovasc Interv. 2011 Mar 1;77(4):510-4. doi: 10.1002/ccd.22734. Epub 2010 Nov 4. PMID 21351225
- [Background] Kandzari DE, Teirstein PS, Kereiakes DJ, Cannon LA, Hearne SE, Kuo HC, Ying SW, Cheong WF, Popma JJ. Procedural effectiveness of a novel 1.20 mm diameter angioplasty catheter: clinical and angiographic outcomes. J Interv Cardiol. 2013 Apr;26(2):131-6. doi: 10.1111/j.1540-8183.2013.12021.x. Epub 2013 Jan 31. PMID 23369084